CLINICAL TRIAL: NCT02991235
Title: Evaluation of the Efficacy and Safety of PRJ212 on Improving the Memory of Patients With Mild Severity Alzheimer's Disease: A 6-month Randomized, Double-blind and Placebo-controlled, Followed by a 6-month Open Label Extension Study
Brief Title: Efficacy and Safety of PRJ212 to Improve the Memory of Patients With Mild Severity Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bioiberica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: BIO-PRJ-2015-01
Record Dates: First submitted 2016-11-29; First posted 2016-12-13 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRJ212 (Experimental): PRJ212 is a nutritional product with active food ingredients.
  Interventions: Dietary Supplement: PRJ212
- Placebo (Placebo Comparator): Placebo is like PRJ212 without active food ingredients.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: PRJ212 — 6 capsules of study product will be taken daily and orally.
  Arms: PRJ212
Dietary Supplement: Placebo — 6 capsules of study product will be taken daily and orally.
  Arms: Placebo

SUMMARY:
A 6-month randomized, double-blind and placebo-controlled, followed by a 6-month open label extension study.

DETAILED DESCRIPTION:
Men and women from 60 to 85 years old with diagnosis of mild severity Alzheimer's disease, according to the diagnostic criteria established by the National Institute of Neurological and Communicative Disorders and Stroke and Alzheimer's Disease and Related Disorders Associations (NINCDS-ADRDA).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 60 to 85 years.
* Patients with a diagnosis of probable or possible Alzheimer's disease according to the NINCDS-ADRDA.
* Patients with mild Alzheimer's disease according to MMSE.
* Patients with ability to ingest oral medication.
* Patients able to undergo a MRI.

Exclusion Criteria:

* Pregnant or breastfeeding women or planning a pregnancy during the study.
* Patients and caregivers unwilling or unable to perform cognitive testing.
* Patients taking part in an interventional clinical trial.
* Patients who have a risk of non-compliance to the study procedures.
* Patients with clinical or significant laboratory abnormalities.
* Patients treated with concomitant treatment or food supplements which could interfere with evaluation criteria.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of PRJ212 versus placebo on the memory measured by Repeatable Battery for the Assessment of Neuropsychological Status (R-BANS). | Comparison of the R-BANS score, from baseline to 6 months.
Efficacy of PRJ212 versus placebo on the memory measured by Wechsler Memory Scale (WMS). | Comparison of the WMS score, from baseline to 6 months.
Efficacy of PRJ212 versus placebo on the memory measured by memory composite (R-BANS+WMS). | Comparison of the total memory composite score, from baseline to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Martinez, Study Director — Bioiberica, S.A.
Locations (1):
- Fundació ACE, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No